CLINICAL TRIAL: NCT07204249
Title: Glutide for Ending Methamphetamine
Acronym: GEM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director of Substance Use Research, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UG3DA063329 (NIH)
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Methamphetamine-dependence
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be blinded. Study drug or placebo will be prepared by an unblinded clinician. Study drug or placebo will be administered by a blinded clinician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Wegovy) (Experimental)
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Semaglutide
  Arms: Semaglutide (Wegovy)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
GEM is a two-phase study to evaluate the use of semaglutide (Wegovy) for the treatment of methamphetamine use disorder (MeUD).

The first phase is a pilot study, which will be an open-label, single-arm pilot study of 25 participants. Participants will receive Wegovy over a 12-week treatment period, with a subsequent follow-up visit at week 20. This phase will evaluate the feasibility, acceptability, and preliminary efficacy of Wegovy for MeUD.

The second phase will be a phase IIb randomized-controlled trial to determine the efficacy of Wegovy in treating MeUD. This trial will be similar to the pilot with randomization to Wegovy or placebo and blinding of group assignment. The trial will enroll 162 participants across two sites.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Ability to provide informed consent before any study-related activity, willing to comply with all study procedures, and be available for the duration of the study,
2. Age 18 - 65 years inclusive,
3. Moderate to severe Methamphetamine Use Disorder by Structured Clinical Interview for DSM Disorders (SCID),
4. Self-reported methamphetamine use ≥15 days out of the past 30,
5. Methamphetamine-positive urine during screening and run-in period,
6. Interested in stopping or reducing meth use,
7. BMI ≥ 25kg/m2,
8. Have at least 1 centimeter of scalp hair,
9. Agree (if the participant is of child-bearing potential) to use effective contraceptive methods, unless all of the participant's male partner(s) is/are surgically sterile (underwent vasectomy). Acceptable contraceptives include oral contraceptives, contraceptive sponge, patch, double barrier (diaphragm/spermicidal or condom/spermicidal), intrauterine contraceptive system, etonogestrel implant, medroxyprogesterone acetate contraceptive injection, complete abstinence from sexual intercourse, and/or hormonal vaginal ring. Contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use. Women of child-bearing potential must provide negative urine pregnancy test prior to randomization.

   Note: A woman is considered fertile (of childbearing potential) following menarche and until becoming postmenopausal unless permanently sterile. Women in the following categories are not considered of childbearing potential: premenarcheal, premenopausal female with one of the following: documented hysterectomy, documented bilateral salpingectomy, documented bilateral oophorectomy. Postmenopausal female is defined as no menses for 12 months without an alternative medical cause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the trial.
10. Be able to provide the names of at least 2 persons who can consistently locate their whereabouts.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Uncontrolled hypertension or systolic BP >160 mmHg and/or diastolic BP >90 mmHg, averaged from three measurements,
2. Resting heart rate greater than 100 bpm at baseline, on at least two measurements,
3. Diabetes (type 1 or 2), hemoglobin A1c ≥ 6.5 at screening, or history of diabetic ketoacidosis,
4. History or current hypoglycemia (blood glucose <70 mg/dL),
5. History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed.
6. History of heart failure or severe gastrointestinal disease (including acute or chronic pancreatitis, any gastric emptying disorder, gallbladder disease; any gastric resection),
7. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia 2A or 2B,
8. Impaired renal function (estimated GFR <60 ml/min),
9. Lipase, amylase, direct (conjugated) bilirubin, or alkaline phosphatase (ALP) 1.5 times the upper limit of normal, or ALT or AST more than 2.5 times the upper limit of normal,
10. Calcitonin value equal to or above 50 ng/L,
11. History of retinopathy,
12. Women who are currently pregnant, or plan to become pregnant, or lactating, or of childbearing potential and are not using medically accepted forms of contraception (see inclusion criterion 9 regarding medically accepted forms of contraception).
13. Acute or chronic illnesses likely to result in hospitalization or death during trial participation,
14. Plan to have all hair removed or chemically treat hair during study,

Psychiatric/Substance Use Exclusions:

1. Moderate to severe opioid, cocaine, or alcohol use disorder,
2. Current non-drug-induced psychotic disorder by Structured Clinical Interview for DSM Disorders (SCID),
3. History of a suicide attempt or past 30-day suicidal ideation,
4. Have any psychiatric illness or condition which in the opinion of the PI and/or the Study Physician would preclude safe and/or successful completion of the study,

Weight-related exclusions:

1. Uncontrolled thyroid disease,

Medication-related exclusions:

1. Past 30 day use of sulfonylureas, insulin and insulin products, or medication used for weight management (e.g., orlistat, naltrexone-bupropion, liraglutide, semaglutide, tirzepatide, phentermine, topiramate, benzhetamine, diethylpropion, phendimetrazine).
2. Prior use of or known hypersensitivity to any GLP-1 agonist,
3. Any otherwise not specified concomitant medication that could compromise participant safety or treatment in the opinion of the Study Physician and/or the PIs,

General exclusions:

1. Current, anticipated, or pending enrollment in another addiction treatment program and/or research study that could potentially affect participant safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
2. Planning to leave the area during the trial,
3. Surgery scheduled during the trial, except for minor surgical procedures that, in the opinion of the PI and/or the Study Physician, will not require general anesthesia with the risk of aspiration,
4. Unable to communicate (read, write, and speak) fluently in English, OR
5. Any other condition that, in the PI's judgment, interferes with safe study participation or adherence to study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-02-15 (Estimated); Study Completion 2030-02-15 (Estimated)

PRIMARY OUTCOMES:
Ratio of eligible to enrolled participants | 14 months
  Feasibility of Wegovy for MeUD treatment: Feasibility will be determined by measuring the ratio of eligible to enrolled participants
Proportion of on-time injections | 20 months
  Acceptability of Wegovy for MeUD treatment: Acceptibility of the treatment will be determined by measuring the adherence to available study drug injections (proportion of on-time injections administered)
Past month methamphetamine use at baseline vs. week 12 | 12 weeks
  Reduced methamphetamine use: Signs of reduced methamphetamine use by hair testing or self-report (timeline follow back) for the past four weeks, measured at baseline vs. week 12.
Rate of study-drug discontinuation | 12 weeks
  Safety of Wegovy for MeUD treatment: Safety will be determined by measuring the rate of study-drug discontinuation due to adverse events
Reduced methamphetamine use | 12 weeks
  Reduced methamphetamine use, measured by proportion achieving "response," defined as 3 out of the final 4 urines collected negative for methamphetamine.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT07204249/Prot_SAP_000.pdf